CLINICAL TRIAL: NCT04832009
Title: Reversing Glucose and Lipid-mediated Vascular Dysfunction (REGAL)
Brief Title: Reversing Glucose and Lipid-mediated Vascular Dysfunction
Acronym: REGAL
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Seth Holwerda PhD, Principal Investigator, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 00147066
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Blood Pressure; Hypertension
MeSH Terms: conditions — Hypertension | interventions — Glucose; Injections; soybean oil, phospholipid emulsion; Lipids; Sodium Chloride; Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Comparisons of outcome variables will be made using a mixed model ANOVA.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomized, double-blinded, parallel-design approach study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glucose Infusion (Experimental): Hyperglycemia (glucose infusion) will receive an I.V. Glucose infusion with a co-infusion of ascorbic acid or placebo at your visit 2 and the alternative treatment of ascorbic acid or placebo will be given on the subsequent study visit 3.
  Interventions: Drug: Dextrose 20 % in 500 ML Injection; Drug: Saline; Drug: Ascorbic acid
- Lipid Infusion (Experimental): Hyperlipidemia (lipid infusion) will receive an I.V. Lipid infusion with a co-infusion of ascorbic acid or placebo at your visit 2 and the alternative treatment of ascorbic acid or placebo will be given on the subsequent study visit 3.
  Interventions: Drug: Intralipid; Drug: Saline; Drug: Ascorbic acid

INTERVENTIONS:
Drug: Dextrose 20 % in 500 ML Injection — Dextrose (20% intravenous solution) will be obtained from the Investigational Pharmacy located in the KU Clinical Research Center where studies take place. After fasting for at least 8 hours, dextrose will be administered via antecubital vein at a standard rate of 4 mg/kg/min for 2 hours.
  Other Names: Glucose
  Arms: Glucose Infusion
Drug: Intralipid — Intralipid ® 20% will be obtained from the Investigational Pharmacy located in the KU Clinical Research Center where studies take place. After fasting for at least 8 hours, Intralipid ® 20% will be administered via antecubital vein at 0.75 mL/min for 2 hours Increases in circulating markers of oxidative stress peak within 2 hours of Intralipid ® 20% infusion in healthy adults (42). An initial heparin bolus of 1000 UL followed by 200 U/hr infusion will be included to activate endothelial lipoprotein lipase and accelerate hydrolysis of fatty acids.
  Other Names: Lipid
  Arms: Lipid Infusion
Drug: Saline — Saline will be obtained from the Investigational Pharmacy located in the KU Clinical Research Center where studies take place. Will be administered via antecubital vein at 75 to 150 mL/hour for 2 hours.
  Other Names: Placebo
Drug: Ascorbic acid — (ASCOR) will be obtained from the KU Investigational Pharmacy located in the KU Clinical Research Center where studies will take place. A priming bolus of 0.06 g ascorbic acid/kg fat free mass (FFM) dissolved in 100 mL of saline will be infused intravenously at 5 mL/min for 20 minutes, followed immediately by a "drip-infusion" of 0.02 g/kg FFM dissolved in 30 mL of saline administered over 2 hours at 0.5 mL/min. The KU Investigational Pharmacy will randomize ascorbic acid or placebo (saline) for each participant.

SUMMARY:
The purpose of our study is to understand the extent to which the blood vessels are affected by glucose and fat (lipids) in lean healthy adults and if these changes in the blood vessels contribute to the development of high blood pressure.

DETAILED DESCRIPTION:
Hypertension, obesity, and insulin resistance are associated with elevated muscle sympathetic nerve activity (MSNA), which is important for blood pressure regulation. The measurement of MSNA is safely performed in humans using the microneurographic technique that involves recording sympathetic nerve activity projecting to skeletal muscle using a small microelectrode at the peroneal nerve near the knee.

The health of your blood vessels will be tested in this study, in addition to the activity of the nerves that control the blood vessels. The function of the nerves and blood vessels can be diminished by high blood glucose and lipids, and we will test the ability of a well-known antioxidant, ascorbic acid (vitamin C), to restore the function of the nerves and blood vessels.

ELIGIBILITY:
Inclusion Criteria:

* Lean: BMI < 25 kg/m
* Normal insulin sensitivity: (calculation based on fasting glucose and insulin concentrations in blood)
* Middle-aged: 18-79 years
* Blood pressure: < 140 (systolic) and < 90 mmHg (diastolic
* Weight stable (+/- 5 lbs) for the previous 3 months
* Participants must be willing and able to discontinue taking any vitamin C or E supplements or omega-3 fatty acids beginning 2 weeks prior.
* Able and willing to provide written informed consent

Exclusion Criteria:

* Diabetes mellitus Type I or Type II: fasting glucose < 126 mg/dL and/or HbA1c < 6.5%
* Current smoker or History of smoking in the past 3 months.
* Hyperlipidemia: Fasting triglycerides < 250 mg/dL
* Hypertension: >130/80 mmHg
* History of heart disease (e.g., myocardial infarction, stent, heart attack, stroke, heart failure, valvular heart disease, cardiomyopathy)
* History of vascular disease (e.g., bypass, stroke)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Infusion of Ascorbic Acid | Baseline
  The difference in sympathetic-vascular transduction (mmHg) between ascorbic acid and placebo infusion will be taken as a measure of the modulation of SVT by oxidative stress.
Efficacy of Infusion of Ascorbic Acid | 30 minutes
  The difference in sympathetic-vascular transduction (mmHg) between ascorbic acid and placebo infusion will be taken as a measure of the modulation of SVT by oxidative stress.
Efficacy of Infusion of Ascorbic Acid | 60 minutes
  The difference in sympathetic-vascular transduction (mmHg) between ascorbic acid and placebo infusion will be taken as a measure of the modulation of SVT by oxidative stress.
Efficacy of Infusion of Ascorbic Acid | 90 minutes
  The difference in sympathetic-vascular transduction (mmHg) between ascorbic acid and placebo infusion will be taken as a measure of the modulation of SVT by oxidative stress.
Efficacy of Infusion of Ascorbic Acid | 120 minutes
  The difference in sympathetic-vascular transduction (mmHg) between ascorbic acid and placebo infusion will be taken as a measure of the modulation of SVT by oxidative stress.

CONTACTS AND LOCATIONS:
Overall Officials: Seth W. W Holwerda, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No